CLINICAL TRIAL: NCT03217682
Title: Impact of Massage Therapy and Music Therapy on the Quality of Life of Hospice Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria I. Lapid, M.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-002950
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Pain; Anxiety; Depression; Quality of Life
Keywords: Hospice; Palliative Care; Integrative Medicine; Massage Therapy; Music Therapy; Caregivers
MeSH Terms: conditions — Pain; Anxiety Disorders; Depression | interventions — Music Therapy; Massage

STUDY DESIGN:
Intervention Model Description: After the patient has been registered into the study, they will be assigned to either the music therapy or massage therapy cohort. The music therapy cohort will be available to the first 30 patients and 30 caregivers accrued. Upon reaching 60 subjects enrolled, the music therapy cohort will close to accrual and the massage therapy cohort will open to accrual. Once the massage therapy cohort has enrolled 30 patients and 30 caregivers, the massage therapy cohort will close to accrual and the study will be closed to all further accrual.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Music therapy twice a week for two weeks, each session lasting approximately 45 min-1 hr
  Interventions: Other: Music Therapy
- Massage Therapy (Experimental): Massage therapy twice a week for two weeks, each session lasting approximately 45 min-1 hr
  Interventions: Other: Massage Therapy

INTERVENTIONS:
Other: Music Therapy — Music therapy sessions
  Arms: Music Therapy
Other: Massage Therapy — Massage therapy sessions
  Arms: Massage Therapy

SUMMARY:
This is a cohort study where subjects will receive either massage therapy or music therapy interventions to evaluate their impact on hospice patients.

DETAILED DESCRIPTION:
There is growing evidence that integrative therapies such as massage therapy and music therapy can be effective therapeutic tools for relief of pain and non-pain symptoms in hospice and palliative care patients. Massage and music therapies can provide comfort, relaxation, and improve quality of life for patients. The investigator's primary aim is to compare the effects of massage and music therapies on the quality of life of hospice patients. The overall goal is to further improve pain, depression, anxiety, and poor well-being or quality of life in hospice patients through the use of integrative therapies, specifically massage and music therapies, as add-on to standard hospice clinical care. Patients will be assigned to either the massage therapy or music therapy cohort. Questionnaires will be utilized before and after each massage or music therapy intervention to quantify symptom and quality of life levels.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently enrolled in Mayo Clinic Hospice
* Age 18 years or older
* ESAS-r scores of 5 or greater on pain, depression, anxiety, or best well-being (clinical assessment by hospice nursing staff)
* Patient or caregiver must be able to participate in brief interviews and complete questionnaires (verbally or physically)

Exclusion Criteria:

* Patients that would not be able to get a massage due to complexity of medical care including complex wound and multiple drains

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Change in Edmonton Symptom Assessment System - Revised | Baseline to 3 weeks
  The primary endpoints are patient pain, depression, anxiety and wellbeing as measured by ESAS-r. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores. The pro-rated AUC for ESAS-r measured pain, depression, anxiety, and wellbeing will all be utilized individually to assess the primary endpoint. The pro-rated AUC will be compared to the assessment score prior to any massage or music therapy. If there is any improvement, the therapy will be considered a success since any improvement will be seen as beneficial.

SECONDARY OUTCOMES:
Change in Edmonton Symptom Assessment System - Revised (Other symptoms) | Baseline to 3 weeks
  Secondary endpoints include all other symptoms (tiredness, drowsiness, nausea, lack of appetite, shortness of breath) as measured by the ESAS-r. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores.
Change in Linear Analogue Self Assessment (LASA) | Baseline to 3 weeks
  Secondary endpoints include symptoms as measured by the LASA (overall quality of life [QOL], mental well-being, physical well-being, emotional well-being, social activity, spiritual well-being, pain frequency, pain severity, fatigue, and social support). LASA items are stand alone, thus no scoring is necessary, but individual LASA items may be transposed so lower scores mean worse symptoms and higher scores mean less symptoms. This will allow consistency and thus easier data interpretation. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome.
Change in Patient Health Questionnaire for Depression and Anxiety (PHQ-4) | Baseline to 3 weeks
  Secondary endpoints include depression and anxiety symptoms as measured by the PHQ-4. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome.
Change in Pearlin role overload measure (ROM) | Baseline to 3 weeks
  Secondary endpoints include caregiver stress as measured by the ROM. Pro-rated area under the curve (AUC) statistics will be calculated for all individual items and total scores. Similar analysis will be conducted for all other endpoints as was conducted for the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lapid, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials